CLINICAL TRIAL: NCT07355244
Title: The Effect of Self-Affirmation Skills on Pain, Depression, Anxiety, and Stress in Patients Undergoing Mastectomy: A Randomized Controlled Trial
Brief Title: Self-Affirmation Intervention After Mastectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, BARIŞ ÖZDERE, Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 222391
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Breast Neoplasms; Mastectomy; Lymphedema; Pain; Depression; Stress, Psychological
Keywords: Mastectomy; Breast Cancer; Stress; Anxiety; Depression
MeSH Terms: conditions — Breast Neoplasms; Lymphedema; Pain; Depression; Stress, Psychological; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model with two arms: an intervention group and a control group. Participants will be randomly assigned to groups using block randomization via a computer-based system (randomizer.org). The intervention group will receive a structured self-affirmation audio recording with calming background sounds, while the control group will receive standard care without additional intervention. The study is open-label, as masking is not feasible due to the nature of the behavioral intervention.
Masking Description: This study is open-label. Masking was not feasible due to the nature of the behavioral intervention (audio recording of self-affirmation statements). Both participants and investigators were aware of group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Standard Care) (No Intervention): Participants in the control arm will receive standard postoperative care according to hospital protocols. No additional behavioral or psychological intervention will be administered.
- Intervention Group (Self-Affirmation Audio) (Experimental): Participants in the intervention arm will receive a behavioral intervention consisting of an audio recording of positive self-affirmation statements accompanied by calming background sounds (birds chirping and flowing water). The recording lasts approximately 5 minutes and 40 seconds and will be delivered via an MP3 player and headphones. Patients will be instructed to listen to the recording at least once daily during the postoperative period, with encouragement to listen more frequently if desired.
  Interventions: Behavioral: Positive Self-Affirmation Audio with Calming Background Sounds

INTERVENTIONS:
Behavioral: Positive Self-Affirmation Audio with Calming Background Sounds — Participants in the intervention arm will receive a behavioral intervention consisting of an audio recording of positive self-affirmation statements accompanied by calming background sounds (birds chirping and flowing water). The recording lasts approximately 5 minutes and 40 seconds and will be delivered via an MP3 player and headphones. Patients will be instructed to listen to the recording at least once daily during the postoperative period, with encouragement to listen more frequently if desired.
  Arms: Intervention Group (Self-Affirmation Audio)

SUMMARY:
This randomized controlled trial aims to evaluate the effect of a structured self-affirmation intervention on pain, depression, anxiety, and stress levels in patients undergoing mastectomy. The study will be conducted in two parallel groups, with the intervention group listening to an audio recording of positive self-affirmation statements. Primary outcomes will be assessed using the Visual Analog Scale and the Depression Anxiety Stress Scale (DASS-21). The goal is to provide evidence-based strategies to reduce psychosocial burden after mastectomy.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to evaluate the effect of a structured self-affirmation intervention on pain, depression, anxiety, and stress levels in patients undergoing mastectomy. Breast cancer is the most commonly diagnosed cancer among women worldwide, and mastectomy, a standard surgical treatment, often results in significant physical and psychosocial consequences. The loss of a breast, perceived as a symbolic part of femininity, can severely impact body image and self-esteem, leading to psychological distress symptoms such as depression, anxiety, and stress, as well as chronic pain. These adverse effects not only reduce quality of life but also negatively influence treatment adherence and long-term survival.

In this study, participants in the intervention group will listen to an audio recording containing positive self-affirmation statements accompanied by soothing background sounds such as birds chirping and flowing water. The recording, prepared by a certified practitioner, lasts approximately 5 minutes and 40 seconds. Patients will be instructed to listen to the recording at least once daily, with encouragement to listen more frequently if desired. The control group will receive standard care without any additional intervention. Primary outcomes will be assessed using the Visual Analog Scale (VAS) for pain and the Depression Anxiety Stress Scale (DASS-21) for psychological distress. The ultimate goal of this trial is to develop an evidence-based nursing and psychosocial support protocol that can be integrated into postoperative care to reduce psychosocial burden and improve well-being in mastectomy patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Female patients who have undergone mastectomy surgery
* Able to speak and understand Turkish
* Provides informed consent and agrees to participate voluntarily

Exclusion Criteria:

* Diagnosed psychiatric disorder
* Hearing impairment that prevents listening to the audio intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Baseline (preoperative, T0), postoperative day 1 (T1), postoperative day 3 (T2, before discharge), and day 10 follow-up (T3).
  Measured using the Visual Analog Scale (VAS), scored from 0 (no pain) to 10 (worst pain).
Depression, Anxiety, and Stress (DASS-21 subscales) | T0 (preoperative baseline), T1 (post-op day 1), T2 (post-op day 3, before discharge), T3 (post-op day 10 follow-up).
  Assessed using the DASS-21 (validated Turkish version), a 21-item instrument with three subscales (depression, anxiety, stress), Likert 0-3; reliability previously reported (Cronbach's α ~0.88 in this study)

SECONDARY OUTCOMES:
Intervention adherence (daily listening frequency) | From T0 training through T3 (daily tracking until day 10 post-op).
  Number of completed listening sessions per day recorded on the "Listening Adherence Log"; minimum once daily recommended during hospitalization and until day 10 post-op.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality and ethical considerations.